CLINICAL TRIAL: NCT01530958
Title: The Kidney Awareness Registry and Education Study
Brief Title: Kidney Awareness Registry and Education
Acronym: KARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 11-07399; 1R34DK093992-01 (NIH)
Record Dates: First submitted 2012-02-07; First posted 2012-02-10 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: CKD; Automated Telephone Self Management; Registry; CKD awareness; Self efficacy
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ATSM + Health Coach and CKD Registry (Experimental)
  Interventions: Behavioral: CKD Registry; Behavioral: ATSM + Health Coach
- CKD Registry (Active Comparator)
  Interventions: Behavioral: CKD Registry
- ATSM + Health Coach (Active Comparator)
  Interventions: Behavioral: ATSM + Health Coach
- Usual Care (no interventions) (Placebo Comparator)
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: CKD Registry — Primary care providers (PCPs) will have access to a Chronic Kidney Disease (CKD) registry for patient care. The registry will:
  * identify patients with CKD
  * notify PCPs of a patients' CKD status
  * provide PCP outreach with NKDEP guidelines and patient educational materials
  Arms: ATSM + Health Coach and CKD Registry; CKD Registry
Behavioral: ATSM + Health Coach — Patients with CKD will participate in an Automated Telephone Self Management (ATSM) program, which blends automated phone calls with live targeted call-backs from a health coach. Patients will receive bi-weekly automated calls for 52 weeks in their native language, consisting of pre-recorded queries pertaining to CKD management, preventive services, and lifestyle changes. Patients will interact with the system using a touch-tone keypad; Out-of-range values or invalid responses will prompt a live call-back within 24-48 hours by a health coach.
  Arms: ATSM + Health Coach; ATSM + Health Coach and CKD Registry
Behavioral: Usual care — Primary care providers will manage their patients with CKD per usual care.
  Patients will receive usual care.
  Arms: Usual Care (no interventions)

SUMMARY:
The purpose of this study is to evaluate the feasibility and acceptability of two different interventions aimed at improving health outcomes among patients with chronic kidney disease (CKD), who are at high risk of CKD progression. Specifically, this study will examine how best to implement a provider-level intervention (access to a CKD-registry) and a patient-oriented intervention (automated telephone self-management (ATSM) + health coach) on patient health outcomes, with a 2x2 factorial design.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD (defined as estimated Glomerular Filtration Rate < 60ml/min/1.73m2 or proteinuria consistently over 3 months) who speak English, Spanish or Cantonese and have a primary care provider

Exclusion Criteria:

* Kidney transplant recipients; pregnant women; individuals with an eGFR <15 ml/min/1.73 m2; prevalent dementia; impaired cognition or severe mental illness; expected life expectancy <6 months; no phone access; self-reported hearing impairment; severe visual impairment preventing use of a touch-tone telephone keypad; and non-study language

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure measurement at baseline and at one year follow-up | Baseline and one year follow-up
  Blood pressure will be measured at baseline and also at the follow-up visit at one year

SECONDARY OUTCOMES:
Change in CKD awareness, functional status, and symptoms at baseline and at one year follow-up | Baseline and one year follow-up
  CKD awareness, functional status, and symptoms will be measured at baseline and also at the follow-up visit at one year. Assessments will be made by standardized phone calls throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Powe, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco Department of Public Health, San Francisco, California
  - San Francisco General Hospital, San Francisco, California

IPD SHARING:
Plan to Share IPD: Undecided
Data may be available upon contact of study PI.

REFERENCES:
- [Derived] Campbell ZC, Dawson JK, Kirkendall SM, McCaffery KJ, Jansen J, Campbell KL, Lee VW, Webster AC. Interventions for improving health literacy in people with chronic kidney disease. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD012026. doi: 10.1002/14651858.CD012026.pub2. PMID 36472416
- [Derived] Machen L, Handley MA, Powe N, Tuot D. Engagement With a Health Information Technology-Augmented Self-Management Support Program in a Population With Limited English Proficiency: Observational Study. JMIR Mhealth Uhealth. 2021 May 11;9(5):e24520. doi: 10.2196/24520. PMID 33973868
- [Derived] Tuot DS, Rubinsky AD, Velasquez A, McCulloch CE, Schillinger D, Handley MA, Hsu CY, Powe NR. Interventions to Improve Blood Pressure Control Among Socioeconomically Disadvantaged Patients With CKD: Kidney Awareness Registry and Education Pilot Randomized Controlled Trial. Kidney Med. 2019 Aug 30;1(5):242-252. doi: 10.1016/j.xkme.2019.07.004. eCollection 2019 Sep-Oct. PMID 32734204
- [Derived] Tuot DS, Velasquez A, McCulloch CE, Banerjee T, Zhu Y, Hsu CY, Handley M, Schillinger D, Powe NR. The Kidney Awareness Registry and Education (KARE) study: protocol of a randomized controlled trial to enhance provider and patient engagement with chronic kidney disease. BMC Nephrol. 2015 Oct 22;16:166. doi: 10.1186/s12882-015-0168-4. PMID 26494562